CLINICAL TRIAL: NCT05679323
Title: The Effect of Early Versus Traditional Hospital Discharge on Activities of Daily Livingfor Women Undergoing Elective Cesarean Section.An Observational Cohort Study.
Brief Title: Evaluation of Early Discharge After Cesarean Section
Status: Completed | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Elmaraghy, Lecturer, Ain Shams Maternity Hospital
Other Study IDs: 8
Record Dates: First submitted 2022-12-22; First posted 2023-01-11 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Early Discharge of Patients After Cesarean Section
MeSH Terms: interventions — Activities of Daily Living

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early discharge: Patients who will be discharged 24 hours after cesarean section
  Interventions: Other: KATZ index of independence in activities of daily living
- Traditional discharge: Patients who will be discharged 48 hours after cesarean section
  Interventions: Other: KATZ index of independence in activities of daily living

INTERVENTIONS:
Other: KATZ index of independence in activities of daily living — KATZ index measures self-care tasks using a dichotomous rating (dependent-0/independent-1) including; bathing, dressing, toileting, transferring to and from a chair, maintaining continence, and feeding. Six points are considered independent and 0 points are considered fully dependent. Assessment of each patient is made through a phone call at day 1, 3 and 5 after discharge

SUMMARY:
The rate of cesarean delivery is increasing, in developing countries, its rate ranges from 13 to 47% of all cases of delivery. This huge volume of cesarean deliveries has a great financial burden on the healthcare system. Rising hospital costs have led to the implementation of an early discharge policy after surgeries.

DETAILED DESCRIPTION:
Cesarean section (CS) is the most commonly performed surgical procedure worldwide that effectively prevents maternal and newborn mortality when used for medically indicated reasons. Compared with vaginal delivery, however, the procedure is associated with a higher risk of various maternal complications, such as maternal infection and subsequent pregnancy complications, and a higher likelihood of re-hospitalization within six weeks of delivery. Furthermore, the likelihood of maternal morbidity increases for mothers who repeatedly undergo cesarean delivery. CS typically implies a hospital stay for two to three days, whereas parous women are often discharged within a few hours after an uncomplicated vaginal birth. However, the period after CS includes recovery from surgery as well as adapting to motherhood.

According to World Health Organization, the cesarean section rate will increase to 28.5% of total live births by the year 2030. This huge volume of cesarean deliveries and increasing cesarean section rate has an incremental burden on the healthcare system, leading to higher bed occupancy and financial pressure on the patients and health facilities. Postpartum stay at hospitals is steadily declining in the UK and other countries due to cost savings. Rising hospital costs are one of the factors in early discharge.

According to The American College of midwifery and gynecology, earlier discharge is a choice if the baby is ready to go home, though, the mother should have basic requirements such as normal blood pressure, no symptoms of infection, and adequate pain control. Also, the National institute for health and care excellence (NICE) guidelines recommend "women who are recovering well, are apyrexial and do not have complications following Caesarean Section should be offered early discharge (after 24 hours) from the hospital and follow up at home.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≤ 35 kg/m2
* Gestational age at delivery from 37 0/7 to 42 0/7 weeks of gestation
* Uncomplicated pregnancy
* Cesarean section under spinal anesthesia with no intra-operative complications
* Uneventful postoperative course

Exclusion Criteria:

* Complicated pregnancy (Multiple pregnancies, Polyhydramions, Abnormal placenta, Premature rupture of membranes).
* Medical disorders (diabetes, hypertension, cardiac, renal, endocrinological disorders).

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women admitted to Ain Shams University Maternity Hospital scheduled for elective lower-segment cesarean section
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Activities of daily living | The first week after cesarean section
  Objective assessment is made by the KATZ index of independence of activities of daily living. The Katz index measures six self-care tasks including; bathing, dressing, toileting, transferring, maintaining continence, and feeding using a dichotomous rating (dependent-0/independent-1). Six points are considered independent and 0 points are considered fully dependent

SECONDARY OUTCOMES:
Wound assessment | First postpartum visit 1 week after the cesarean section
  Assessment of the wound by the Southampton wound scoring system will take place 1 week after the cesarean section. It categorizes wound complications on a grade from 0 to V, with the latter being deep or severe wound infection.
Return to normal bowel activities | First 48 hours after cesarean section
  Passage of flatus and stool after the cesarean section
initiation of successful breast feeding | First postpartum visit 1 week after the cesarean section
  Start of lactation
Neonatal readmission | First postpartum visit 1 week after the cesarean section
  The rate of neonatal admission and the reason will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M ElMaraghy, MD, Principal Investigator — Ainshams university maternity hospital; Ahmed H Naguib, MD, Study Director — Ainshams university maternity hospital; Ahmed M Fahim Hemaid, MD, Study Chair — Ainshams university maternity hospital
Locations (1):
- AinShams university maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fikrie A, Zeleke R, Bekele H, Seyoum W, Hailu D, Wayessa ZJ, Tufa G, Utura T, Matie M, Oda GD. Time-to-recovery after cesarean section delivery among women who gave birth through cesarean section at Hawassa University Comprehensive Specialized Hospital, South Ethiopia: A prospective cohort study. PLOS Glob Public Health. 2022 Oct 5;2(10):e0000696. doi: 10.1371/journal.pgph.0000696. eCollection 2022. PMID 36962571
- [Background] Sakai-Bizmark R, Ross MG, Estevez D, Bedel LEM, Marr EH, Tsugawa Y. Evaluation of Hospital Cesarean Delivery-Related Profits and Rates in the United States. JAMA Netw Open. 2021 Mar 1;4(3):e212235. doi: 10.1001/jamanetworkopen.2021.2235. PMID 33739430
- [Background] Kruse AR, Lauszus FF, Forman A, Kesmodel US, Rugaard MB, Knudsen RK, Persson EK, Uldbjerg N, Sundtoft IB. Effect of early discharge after planned cesarean section on recovery and parental sense of security. A randomized clinical trial. Acta Obstet Gynecol Scand. 2021 May;100(5):955-963. doi: 10.1111/aogs.14041. Epub 2020 Dec 25. PMID 33179268
- [Background] 4- Gupta S, Gupta A, Baghel AS, Sharma K, Choudhary S, Choudhary V. Enhanced recovery after cesarean protocol versus traditional protocol in elective cesarean section: A prospective observational study. J Obstet Anaesth Crit Care 2022;12:28-33
- [Background] Ghaffari P, Vanda R, Aramesh S, Jamali L, Bazarganipour F, Ghatee MA. Hospital discharge on the first compared with the second day after a planned cesarean delivery had equivalent maternal postpartum outcomes: a randomized single-blind controlled clinical trial. BMC Pregnancy Childbirth. 2021 Jun 30;21(1):466. doi: 10.1186/s12884-021-03873-8. PMID 34193059
- [Background] 6- Trikha A, Kaur M. Enhanced recovery after surgery in obstetric patients - Are we ready?. J Obstet Anaesth Crit Care 2020;10:1-3